CLINICAL TRIAL: NCT07029633
Title: Effect of Cartoon and Storytelling on the Children's Fear and Anxiety Levels During Inhalation Therapy With Nebulizer in Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Sibel Serap Ceylan, Associate professor, PhD, RN, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PamU
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Distraction Methods; Child
Keywords: anxiety; child; fear; cartoon; storytelling
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: randomized controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): To reduce fear and anxiety in the children in this group, the storytelling method was used by the parents during the nebulizer treatments.
  Interventions: Other: storytelling
- Group 2 (Experimental): During nebulizer treatments, children in this group collaboratively chose cartoons on YouTube with their parents and watched them on phones using the hospital's internet.
  Interventions: Other: cartoon
- Group 3 (No Intervention): No intervention was performed on the children in the control group to reduce fear and anxiety related to inhalation therapy with a nebulizer.

INTERVENTIONS:
Other: storytelling — to distract telling a story
  Arms: Group 1
Other: cartoon — to distract watching a cartoon
  Arms: Group 2

SUMMARY:
Inhalation therapy with a nebulizer is a non-invasive and easy-to-use technology. However, the use of masks and the loud, unpleasant sound of the nebulizer can cause fear and anxiety in children. For nebulizer inhalation therapy to be effective, it is important to reduce children's fear and anxiety and to increase their compliance with treatment. Simple and inexpensive distraction methods can be used to achieve this. The results show that cartoon and storytelling methods reduce fear and anxiety in children undergoing inhalation therapy with the nebulizer.

DETAILED DESCRIPTION:
This study aimed to evaluate the impact of cartoons and storytelling during nebulizer inhalation treatment on procedure-related fear and anxiety in children. This randomized controlled study employed a 3-arm parallel design with 99 children aged 5-8 receiving nebulizer therapy in the pediatric emergency department. Groups 1 and 2 served as the experimental groups, while Group 3 acted as the control group, with no intervention addressing fear and anxiety. Group 1 utilized storytelling as a distraction, while Group 2 watched cartoons. Data were collected using the Descriptive Characteristics Form, the Child Follow-Up Form, the Children's Anxiety Meter-State, and the Child Fear Scale.

In the study, parental presence was ensured during the procedure in all groups. For this reason, parents were informed, and their questions about inhalation treatment with nebulizers were answered before data collection to reduce parents' stress and anxiety in all groups and to prevent children from being affected by their parents' emotional situation. The parents were seated in a comfortable chair beside the children's bed.

Before the inhalation treatment with a nebulizer, the procedure was explained to the child according to the child's developmental level, the fear and anxiety levels of the children were evaluated, and their cardiorespiratory rates were measured. Then, inhalation therapy with a nebulizer was started. During the procedure, children's anxiety levels, crying situations, and cardiorespiratory rates were measured. After the procedure, the nebulizer was turned off, the mask was removed, and their faces were cleaned. The children's fear and anxiety levels were evaluated for the last time, and their cardiorespiratory rates were measured. The duration of the inhalation treatment was approximately 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

Children between 5 and 8 years old, who received inhalation therapy with a nebulizer for the first time, had no communication problems, and gave consent were included in the study.

Exclusion Criteria:

Children who had vision, hearing, and comprehension problems, mental and neurological diseases, life-threatening diseases, those who used any medication with sedative effects, or those who refused interventions during nebule treatment were not included in the study.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 99 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
fear level | 15-30 minute
  The Child Fear Scale (CFS) was used children's fear level
anxiety level | 15-30 minute
  To determite anxiety level of children The Children's Anxiety Meter-State (CAM-S) was used.
crying duration | 15-30 minute
  The crying duration of the children during the procedure was measured and recorded by the researchers with a stopwatch.
Cardiorespiratory rates: | 15-30 minute
  Children's respiration rate was measured by observation, pulse rate and SPO2 levels were measured by finger pulse oximeter.

CONTACTS AND LOCATIONS:
Locations (1):
- Sibel Serap Ceylan, Denizli, Pamukkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided